CLINICAL TRIAL: NCT03693053
Title: Assessment of the Level of Precariousness in a Population of Patients With Symptomatic Peripheral Arterial Disease.
Brief Title: Socioeconomic Deprivation and Peripheral Arterial Disease
Acronym: PRECAR
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.212; 2017-A02063-50 (Other: ID RCB)
Record Dates: First submitted 2018-07-31; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Atherosclerosis is a systemic disease that affects coronary, cerebral, and lower-extremity arteries. Peripheral artery disease (PAD) is the manifestation of atherosclerosis in the legs. Three different stages can be found: asymptomatic stage (stage 1), exercise ischemia stage (stage 2) and rest ischemia stage (stage 3). The risk factors for PAD are similar to those for coronary artery disease (CAD) and cerebrovascular disease (CBVD), like high blood pressure, diabetes, smoking, dyslipidemia and obesity. But cigarette smoking is the single most important risk factor for the development and progression of PAD.

PAD is a serious illness and an important predictor of cardiovascular disease with major medico-economic consequences.

A low socioeconomic status (SES) is associated with higher cardiovascular mortality and morbidity. In these vulnerable populations, there is an increase in the prevalence of cardiovascular risk factors, particularly for smoking.

The main objective of this study was to assess the level of precariousness in patients with symptomatic PAD and compare it to the level of precariousness in the general population.

Patients were recruited from vascular medicine and surgery department of Grenoble university hospital or therapeutic education outpatient consultation.

The analysis of socio-economic and environmental data resulted in:

- EPICES score: (Evaluation of the Deprivation and Inequalities of Health in Healthcare Centers score). The EPICES score is a quick and validated questionnaire to assess precariousness at the individual level, developed by considering all the material and psychosocial dimensions of precariousness.

Precariousness, according to the EPICES score, in the general population is estimated at 40%.

- INSEE parameters. The investigators completed the EPICES score with more traditional indicators derived from The National Institute of Statistics and Economic Studies (INSEE) collects, analyses and disseminates information on the French economy and society. The investigators collected the level of education and professional practice based on the nomenclature of socio-professional categories defined by INSEE.

Cardiovascular risk factors were also collected to measure the links between the level of precariousness and cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* Age 18 years or older,
* Symptomatic PAD (stage 2 or 3)

Exclusion Criteria:

* Pregnant woman
* Person under administrative or judicial supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients were recruited from
  * Vascular medicine and surgery department of Grenoble university hospital
  * Or therapeutic education consultation. These consultations took place in Grenoble reference center of therapeutic education CREPvAL Granted as part of education program: "On the move! Better understand and better live your PAD".
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Level of precariousness in patients with symptomatic PAD | one day
  The level of precariousness is measured by EPICES score : It consists of 11 items related to isolation, health insurance status, economic status, social support and leisure activity. For each item, a binary response Yes/No is expected from the patient. The total score ranges from 0 to 100, from lack to the highest social deprivation. Patients were considered precarious if their score is superior to threshold of 30.

SECONDARY OUTCOMES:
Level of precariousness by EPICES score between stage 2 and stage 3 of symptomatic PAD. | one day
  Stade 2 : exercise ischemia stage Stade 3 : rest ischemia stage
Links between the level of precariousness by EPICES score and cardiovascular risk factors. | one day
  Cardiovascular risk factors were:
  Hypertension was defined as a systolic blood pressure of 140 mm Hg or higher, or a diastolic blood pressure of 90 mm Hg or higher, or current use of antihypertensive drugs.
  Hypercholesterolemia was defined as LDL cholesterol levels of 0,7 g/l or higher or current use statin.
  Subjects were considered to have diabetes mellitus if they reported a physician diagnosis of diabetes mellitus, were taking prescription medications for diabetes mellitus (either insulin or oral agents).
  Subjects were classified into groups of current smokers, former smokers (smoking cessation for more than 9 months) and non-smokers.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Grenoble, Isere, France

IPD SHARING:
Plan to Share IPD: No